CLINICAL TRIAL: NCT05930639
Title: The Effect of Care Bundle Applied to Patients Undergoing Bariatric Surgery on Surgical Site ınfection and Comfort
Brief Title: The Effect of the Care Bundle to be Applied to Obesity Surgery Patients on Surgical Site Infection and Patient Comfort
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Malatya Turgut Ozal University (Other)
Responsible Party: Principal Investigator, Hatice ÇAKIR, Research Assistant, Malatya Turgut Ozal University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 2022-07-22/30
Record Dates: First submitted 2023-06-22; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Bariatric Surgery Candidate
Keywords: Surgical Site Infection; Bariatric Surgery; Care bundle; prevention package
MeSH Terms: conditions — Surgical Wound Infection | interventions — Patient Care Bundles

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Surgical Site Infection (SSI) prevention package; Identification of risk factors (Experimental): Risk factors of the individual created in line with the literature; Advanced age, history of skin or soft tissue infection, DM, alcohol addiction, smoking, preoperative albumin <3.5 mg/dl, total bilirubin>1.0 mg/dl, immunosuppression, long postoperative stay, long preoperative stay, high BMI,ASA score > II,preoperative low Hgb level.
  Risk factors associated with the surgical procedure; Presence of drain, prolongation of surgery time, preoperative skin preparation, blood transfusion, non-sterile equipment, insufficient ventilation, heavy operating room traffic, insufficient hemostasis.
  Participants will be evaluated in terms of these risks.
  Interventions: Other: Surgical Site Infection (SSI) prevention package
- Surgical Site Infection (SSI) prevention package; Antibiotic prophylaxis (Experimental): determined antibiotic (active ingredient: imipenem cilastatin sodium)
  Interventions: Other: Surgical Site Infection (SSI) prevention package
- Surgical Site Infection (SSI) prevention package;achieving and maintaining normothermia (Experimental): Body temperature will be recorded with an infrared thermometer. The patient will be warmed with various passive heating techniques before and after the operation. To prevent hypothermia, the operating room ambient temperature will be kept in the range of 23-26°C.
  Interventions: Other: Surgical Site Infection (SSI) prevention package
- Surgical Site Infection (SSI) prevention package; maintenance of normoglycemia (Experimental): In the 2017 guidelines, perioperative glycemic control with a blood glucose level of <200 mg/dL is recommended for patients with and without DM. Ideal blood glucose control should provide good glycemic control with a minimal incidence of hypoglycemia.
  Interventions: Other: Surgical Site Infection (SSI) prevention package
- Surgical Site Infection (SSI) prevention package;patient education (Experimental): SSI definition, SSI signs and symptoms, Hand hygiene, smoking, hair removal in the operation area, shower and bath before surgery. Conditions that require hospitalization, factors affecting wound healing, wound care, control time and who should be contacted will be discussed.
  Interventions: Other: Surgical Site Infection (SSI) prevention package
- control group (No Intervention): Antibiotic prophylaxis is applied to both groups. In the clinic where the study will be conducted, the blood glucose level of patients with a diagnosis of DM is controlled (5 measurements per day). All patients are fasted after 21.00 in the evening. The blood glucose levels of patients without a diagnosis of DM are not routinely checked. The body temperature of the patients is not monitored intraoperatively. No extra intervention is applied to maintain normothermia in the clinic and operating room.
  There is no training on prevention of infection. There is no intervention in the control group.

INTERVENTIONS:
Other: Surgical Site Infection (SSI) prevention package — Care package components to be applied to the intervention group; identification of risk factors, antibiotic prophylaxis, normothermia, normoglycemia and patient education.
  Risk factors will be evaluated when the patient is admitted to the clinic. Antibiotics (imipenem + cilastatin sodium) routinely administered by the institution before surgery will be administered in both groups.
  Passive heating methods will be used to maintain body temperature for the first 24 hours after surgery.
  In the perioperative period, the blood glucose level will be kept below 200mg/dl for 48 hours.
  Before the operation and before discharge, the patient is educated about infection prevention measures.
  Other Names: care bundle; care package
  Arms: Surgical Site Infection (SSI) prevention package; Antibiotic prophylaxis; Surgical Site Infection (SSI) prevention package; Identification of risk factors; Surgical Site Infection (SSI) prevention package; maintenance of normoglycemia; Surgical Site Infection (SSI) prevention package;achieving and maintaining normothermia; Surgical Site Infection (SSI) prevention package;patient education

SUMMARY:
One of the most effective treatment methods of obesity is surgery. Bariatric surgery is classified as a clean-contaminated wound. The expected benefit from surgery is weight loss. However, surgical site infection is among the complications. Although many methods are applied to reduce these rates, it is not very possible to reduce them to zero. It is predicted that the incidence of infection will decrease with surgical care packages created from the combination of evidence-based interventions applied.

This study was a randomized controlled trial designed to determine the effect of the Surgical Site Infection (SSI) prevention package on SSI and patient comfort in patients undergoing bariatric surgery.

The questions to be answered by the research are;

* What is the effect of the care package applied to patients undergoing bariatric surgery on surgical site infection?
* What is the effect of the care package applied to patients undergoing bariatric surgery on comfort? .Patients aged 18 and over who have had bariatric surgery (sleeve gastrectomy) will be taken from a private hospital in Kayseri. All surgeries will be performed by the same surgeon. The care package (identification of risk factors, antibiotic prophylaxis, normothermia, normoglycemia and patient education) prepared for the experimental group will be applied. On the 30th day, the patient is called by phone and the surgical site infection findings are questioned.

DETAILED DESCRIPTION:
Surgical Site Infection (SSI) was identified by the Center for Disease Control and Prevention (CDC) as a secondary surgical infection within 30 days after surgery. 2017 Health Service Related Infections Surveillance Network report in Turkey, according to the overall SSI rate is 0.72. A study in the literature found the incidence of as 22.2% after abdominal surgery. SSI has been shown to affect one in about every five patients undergoing abdominal surgery and has an incidence of approximately 20%-25% ' associated with contamination. In a comprehensive study conducted in Turkey, it was determined that SSI was seen in the third row after upper gastrointestinal (GIS) surgery and 47.06% of the patients were diagnosed with SSI after discharge.

In a retrospective study investigating the factors that predispose to SSI in general surgery; American Society of Anesthesiologists (ASA) score, wound classification (clean-contaminated, contaminated and dirty/infected wounds), operation history, prolongation of operation time, hypoalbuminemia, history of Chronic Obstructive Pulmonary Disease were defined as major risk factors for the development of SSI. Preoperative low hemoglobin, history of congestive heart failure, excessive alcohol use, surgery at the previous incision site, presence of existing infection, long preoperative and postoperative hospital stay, obesity, steroid use, preoperative epilation, operative data (surgeon's experience, incision device) , drain use, prosthetic mesh use, intraoperative blood transfusion) are other risk factors that increase the risk of SSI.It is suggested that by determining risk factors to reduce the incidence of SSI, it reduces hospital stay and health spending and decreases morbidity and mortality rates.

Bariatric surgery is an effective and widely used treatment for obese patients. The expected benefit from this surgical treatment is weight loss. In addition, this surgery can lead to the development of complications that have significant effects on morbidity and mortality.The use of antimicrobial prophylaxis for organisms causing SSI is important in bariatric surgery. The purpose of antibiotic prophylaxis is to reduce the bacterial load to a level that can be controlled by host defenses.

İnadvertent Perioperative Hypothermia (IPH) (body temperature below 36 °C) is a risk factor for the development of SSI. In a study investigating the effect of hypothermia on SSI in gastroenterological surgery, hypothermia was found to be associated with a higher incidence of organ/space SSI. IPH can cause prolonged hospital stay, cardiac morbidity, increased blood loss, and many complications such as tissue hypoxia and SSI due to neutrophil dysfunction.The CDC recommends maintaining perioperative normothermia to prevent SSI, and the recommendation is considered as the evidence level category IA. The current guidelines propose to use effective heating methods to maintain normothermia in the perioperative period and to measure the patient's body temperature.

Hyperglycemia is another independent risk factor for SSI. In a retrospective study, it was shown that serum glucose level higher than 110 mg/dL is associated with a gradual increase in post-surgical infection rates, and performing glycemic control in the first 48 hours after surgery reduces SSIs. CDC recommended performing perioperative glycemic control in patients with and without diabetes and use blood glucose target levels below 200 mg/dL.( Category IA - strong recommendation; high to medium quality evidence ). Hyperglycemia is a preventable variable to reduce the incidence of SSI.

Another important factor for SSI prevention is patient education. For this reason, the patient and his family should be trained to prevent proper wound care and SSI. However, the benefit of existing patient education materials is uncertain, and a limited number of patient training materials for SSI prevention were found for patients with bariatric surgery.

The concept of "Care Package" has been brought to the agenda by the American Institute for Healthcare Improvement (IHI) in order to achieve more optimal results by applying the interventions with positive results individually in line with evidence-based approaches. IHI has the criteria for inclusion of an element in the care package; It has identified it as consensus and high acceptance, providing solid evidence for clinical change, with little or no discussion of its activities. Maintenance packages with few and simple items have been determined to have better compliance rates. In a systematic review and meta-analysis study, it was reported that the use of SSI measure packages was estimated to prevent 60% of the incidence of SSI. SSI is a complex problem affected by many factors. SSI reduction strategies are multimodal and take place in a number of environments under the supervision of a large number of providers. Ensuring a high level of compliance with these risk reduction strategies is crucial to the success of SSI mitigation efforts.

In different studies, in which multidisciplinary care packages aimed at preventing SSI were applied, significant reductions were achieved in the long term and the use and development of care packages was recommended. Packages can improve the quality of surgical care for patients by providing a harmonious environment and standardization, effectively reducing the risk of SSI. This improvement in the quality of care may increase the comfort level of patients.The concept of comfort in the nursing discipline is based on meeting the needs and is accepted as a part of quality care.

This study is planned to determine the effect of the SSI prevention package on SSI and patient comfort in patients undergoing bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over
* undergoing sleeve gastrectomy surgery
* who volunteered to participate in the study

Exclusion Criteria:

* under 18 years old
* Surgeries other than sleeve gastrectomy
* not willing to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Surgery Site Infection | The infection will be evaluated in the hospital on the 7th day after surgery. An evaluation will be made by phone call on the 30th day after the operation.
  The Centers for Disease Control and Prevention (CDC) defined SSI as an infection secondary to surgery in the superficial, deep or organ cavity within 30 days of surgery. On the 7th day after surgery, the wound will be observed for infection while the stitches are removed. In the presence of symptoms such as purulent discharge, pain, increased redness, swelling and tenderness in the surgical area within 30 days, they will be referred to a health institution for the detection of SSI

SECONDARY OUTCOMES:
Perianesthesia Comfort Scale | Postoperative 0-1. day
  Perianesthesia Comfort Scale, which consists of 24 items measuring the postoperative comfort level, will be applied.

CONTACTS AND LOCATIONS:
Overall Officials: Meryem YILMAZ, Study Director — SİVAS CUMHURİYET UNIVERSITY; Hatice ÇAKIR, Principal Investigator — Malatya Turgut Ozal University
Locations (2):
- Turkey (Türkiye) (2):
  - Hatice ÇAKIR, Malatya
  - Meryem Yilmaz, Sivas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aga E, Keinan-Boker L, Eithan A, Mais T, Rabinovich A, Nassar F. Surgical site infections after abdominal surgery: incidence and risk factors. A prospective cohort study. Infect Dis (Lond). 2015;47(11):761-7. doi: 10.3109/23744235.2015.1055587. Epub 2015 Jun 26. PMID 26114986
- [Background] Horan TC, Andrus M, Dudeck MA. CDC/NHSN surveillance definition of health care-associated infection and criteria for specific types of infections in the acute care setting. Am J Infect Control. 2008 Jun;36(5):309-32. doi: 10.1016/j.ajic.2008.03.002. No abstract available. PMID 18538699
- [Background] Isik O, Kaya E, Dundar HZ, Sarkut P. Surgical Site Infection: Re-assessment of the Risk Factors. Chirurgia (Bucur). 2015 Sep-Oct;110(5):457-61. PMID 26531790
- [Background] Haridas M, Malangoni MA. Predictive factors for surgical site infection in general surgery. Surgery. 2008 Oct;144(4):496-501; discussion 501-3. doi: 10.1016/j.surg.2008.06.001. PMID 18847631
- [Background] Alkaaki A, Al-Radi OO, Khoja A, Alnawawi A, Alnawawi A, Maghrabi A, Altaf A, Aljiffry M. Surgical site infection following abdominal surgery: a prospective cohort study. Can J Surg. 2019 Apr 1;62(2):111-117. doi: 10.1503/cjs.004818. PMID 30907567
- [Background] Carvalho RLR, Campos CC, Franco LMC, Rocha AM, Ercole FF. Incidence and risk factors for surgical site infection in general surgeries. Rev Lat Am Enfermagem. 2017 Dec 4;25:e2848. doi: 10.1590/1518-8345.1502.2848. PMID 29211190
- [Background] Wang Z, Chen J, Wang P, Jie Z, Jin W, Wang G, Li J, Ren J. Surgical Site Infection After Gastrointestinal Surgery in China: A Multicenter Prospective Study. J Surg Res. 2019 Aug;240:206-218. doi: 10.1016/j.jss.2019.03.017. Epub 2019 Apr 12. PMID 30986636
- [Background] Chopra T, Zhao JJ, Alangaden G, Wood MH, Kaye KS. Preventing surgical site infections after bariatric surgery: value of perioperative antibiotic regimens. Expert Rev Pharmacoecon Outcomes Res. 2010 Jun;10(3):317-28. doi: 10.1586/erp.10.26. PMID 20545596
- [Background] Berrios-Torres SI, Umscheid CA, Bratzler DW, Leas B, Stone EC, Kelz RR, Reinke CE, Morgan S, Solomkin JS, Mazuski JE, Dellinger EP, Itani KMF, Berbari EF, Segreti J, Parvizi J, Blanchard J, Allen G, Kluytmans JAJW, Donlan R, Schecter WP; Healthcare Infection Control Practices Advisory Committee. Centers for Disease Control and Prevention Guideline for the Prevention of Surgical Site Infection, 2017. JAMA Surg. 2017 Aug 1;152(8):784-791. doi: 10.1001/jamasurg.2017.0904. PMID 28467526
- [Background] Tsuchida T, Takesue Y, Ichiki K, Uede T, Nakajima K, Ikeuchi H, Uchino M. Influence of Peri-Operative Hypothermia on Surgical Site Infection in Prolonged Gastroenterological Surgery. Surg Infect (Larchmt). 2016 Oct;17(5):570-6. doi: 10.1089/sur.2015.182. Epub 2016 Mar 30. PMID 27027205
- [Background] Zellmer C, Zimdars P, Parker S, Safdar N. Evaluating the usefulness of patient education materials on surgical site infection: a systematic assessment. Am J Infect Control. 2015 Feb;43(2):167-8. doi: 10.1016/j.ajic.2014.10.020. Epub 2014 Dec 23. PMID 25541334
- [Background] Ban KA, Minei JP, Laronga C, Harbrecht BG, Jensen EH, Fry DE, Itani KM, Dellinger EP, Ko CY, Duane TM. American College of Surgeons and Surgical Infection Society: Surgical Site Infection Guidelines, 2016 Update. J Am Coll Surg. 2017 Jan;224(1):59-74. doi: 10.1016/j.jamcollsurg.2016.10.029. Epub 2016 Nov 30. No abstract available. PMID 27915053
- [Background] Weiser MR, Gonen M, Usiak S, Pottinger T, Samedy P, Patel D, Seo S, Smith JJ, Guillem JG, Temple L, Nash GM, Paty PB, Baldwin-Medsker A, Cheavers CE, Eagan J, Garcia-Aguilar J; Memorial Sloan Kettering Multidisciplinary Surgical-Site Infection Reduction Team. Effectiveness of a multidisciplinary patient care bundle for reducing surgical-site infections. Br J Surg. 2018 Nov;105(12):1680-1687. doi: 10.1002/bjs.10896. Epub 2018 Jul 4. PMID 29974946
- [Derived] Cakir H, Yilmaz M. Impact of a Care Bundle on Surgical Site Infections and Patient Comfort in Bariatric Surgery: A Randomized Prospective Study. Obes Surg. 2025 Sep;35(9):3810-3821. doi: 10.1007/s11695-025-08116-9. Epub 2025 Aug 23. PMID 40848119